CLINICAL TRIAL: NCT03172741
Title: The Effects of Different Medical Marijuana Strains on Motor and Cognitive Function in People With Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Did not pursue study
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Thorsten Rudroff, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-6964H
Record Dates: First submitted 2017-05-25; First posted 2017-06-01 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Cannabis
MeSH Terms: conditions — Multiple Sclerosis; Marijuana Abuse | interventions — Medical Marijuana; nabiximols; Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo group: THC (0%) / CBD (0%) (Placebo Comparator): The matching dose for high THC, high CBD or mixed CBD/THC is a 1 gram placebo cigarette (THC (0%) / CBD (0%)) smoked once per day of for 3 months.
  Interventions: Drug: Placebo
- CBD group:THC (<1%) / CBD (>10%) (Experimental): The dose for the CBD group (THC (<1%) / CBD (>10%)) is 1 gram medical marijuana cigarette smoked once per day for 3 months.
  Interventions: Drug: Medical Marijuana
- THC group: THC (>10%) / CBD (<1%) THC group (Experimental): The dose for the THC group (THC (>10%) / CBD (<1%)) is 1 gram medical marijuana cigarette smoked once per day for 3 months.
  Interventions: Drug: Medical Marijuana
- Mixed group:THC (5-10%) / CBD (5-10%) (Experimental): The dose for the mixed group THC (5-10%) / CBD (5-10%) ) is 1 gram medical marijuana cigarette smoked once per day for 3 months.
  Interventions: Drug: Medical Marijuana

INTERVENTIONS:
Drug: Medical Marijuana — 1-gram marijuana cigarette smoked once per day for 3 months
  Other Names: Cannabis; Tetrahydrocannabinol; Cannabidiol
  Arms: CBD group:THC (<1%) / CBD (>10%); Mixed group:THC (5-10%) / CBD (5-10%); THC group: THC (>10%) / CBD (<1%) THC group
Drug: Placebo — Matching 1 gram placebo cigarette smoked once per day for 3 months
  Arms: Placebo group: THC (0%) / CBD (0%)

SUMMARY:
Over the last two years, the United States has witnessed enormous change concerning the acceptance of marijuana. The number of persons with MS (PwMS) using cannabis to treat their symptoms is expected to rise, and it is important to provide clinicians and PwMS with evidence based information on the safety and effectiveness of marijuana. In addition, scientists need to identify the effects of medical marijuana as the compound action of different cannabinoids, specifically tetrahydrocannabinol (THC) and cannabidiol (CBD). The ratio of CBD to THC may have an important impact on the effects of the marijuana, which in turn may have important implications for the medical benefits. The overarching goal of this study is to advance a better understanding of the potential positive and negative effects associated with different strains of marijuana, using an interventional design. The investigators will examine three strains that differ markedly on THC potency (A. THC <1%, CBD > 10%; B. THC >10%, CBD < 1%; C. THC 510%, CBD 510%) to determine whether the level of THC is associated with differences in motor and cognitive functions in PwMS. One hundred PwMS will be recruited for this project and followed for 3 months following designation to one of three strains of marijuana with different ratios of CBD to THC or a placebo marijuana (THC 0%, CBD 0%). It is hypothesized that the strains with a high CBD to THC ratios will demonstrate the most benefits on measures of motor and cognitive function.

DETAILED DESCRIPTION:
Prospective participants will be recruited from the Integrative Neurophysiology Laboratory's (INPL) participant database, the clinical practice of Dr. William Shaffer, Banner Health, Greeley Colorado, through advertisements in the Colorado and Wyoming Chapter of the National MS Society newsletters, and via the Rocky Mountain MS Newsletter. All experimental procedures will be performed in the INPL (Director: Thorsten Rudroff, PhD, FACSM).

Interested individuals will perform an initial screening via an online questionnaire, hosted by Qualtrics, which has a contract with the College of Health and Human Sciences.

Contact information for the prospective participants will be accessible only to the research staff according to HIPAA regulations. After completion of the online screening form, INPL personnel will contact eligible participants via phone and establish 100 total participants. After participants have been identified, INPL staff will schedule the participants' first visit. Eligibility requirements for this study are: medically diagnosed with MS, 21-74 years of age, and moderate disability (Patient Determined Disease Steps score 2-6). The investigators will recruit people with MS who are planning to use medical marijuana for the first time for the treatment of their symptoms. All participants must have a medical (red) card for medical marijuana use to treat their MS symptoms (such as neuropathic pain and spasticity), or currently be in the process of applying for a red card and be able to provide the prescription from their doctor. Marijuana and placebo cigarettes will be ordered from the NIDA (National Institute on Drug Abuse) Drug Supply Program and stored at a designated room in the Department of Health and Exercise Science (HES) at Colorado State University (CSU).

The experimental protocol for this study consists of one testing session that will be performed four times:

Once before the assignment of marijuana product and then once a month during this 3 month longitudinal study. All experiments will be conducted by research personnel (outcome assessors) who are blinded to product assignment. Prior to each session the clinical trial administrator (CTA) will perform an urine analysis assessment for Δ9-tetrahydrocannabinol (THC) to confirm compliance.

Upon arrival to the Integrative Neurophysiology Lab (INPL) at CSU the investigators will explain the protocol procedures and receive signed informed consent from the participants. All eligible participants will be randomized to a coded treatment group by the CTA. After the urine analysis assessment, they will be given one of the four coded cannabis products. All participants will be asked to smoke one single 1- gram marijuana or placebo cigarette per day (Hart et al. 2010). Because these are newly marijuana users, they will be informed about the practical and legal limitations, including barriers to travelling with the medication.

Participants will be asked to return to the lab biweekly for their next set of dosages of coded intervention, as coded and dispensed by the CTA. By providing the participants with additional intervention doses intervention compliance can be determined at the biweekly visits by the CTA. Participants will also be given a log to track their cannabis product use. It is expected that the testing session (once / month) will last between 2-3 hours.

MONTHLY ASSESSMENTS:

1. Blood draw with sodium heparin at the beginning of the session.
2. Questionnaires: Participants will complete several questionnaires: Fatigue Severity Scale (FSS), Beck's Depression Inventory (BDI), the MS Quality of Life (MSQOL)-54 Instrument, and the MOS Pain Effects Scale (PES).
3. The next task will be a Dual Task (walking task and cognitive task) (Etemadi, 2016). Subjects will continuously walk for 60 seconds at a preferred speed along a 10 m walk way. The walking velocity will be calculated. During the walking task the participants will be required to make mathematical subtractions of 7 from random numbers between 200 to100. Responses will be recorded using a voice recorder. The score will be calculated as: correct response rate (CRR) = response rate per second × % of correct responses. The CRR had acceptable reliability (ICC = 0.61-0.75) in patients with multiple sclerosis (Ghanavati et al. 2014).
4. Participants will perform the MS Functional Composite (MSFC) which consists of a 25 foot walk test (25FWT), the 9 hole peg test (9HPT), and the Paced Auditory Serial Addition Test (PASAT). For the 25FWT participants will be asked to walk 25 feet as quickly, but as safely as possible. This will be performed in an isolated hallway with the length clearly marked. Participants will begin after a short count down and the time it takes to walk 25 feet will be measured with a handheld stop watch. Two trials of the 25FWT will be performed and INPL staff will walk alongside the participants to minimize the risk of falling. Next, the 9HPT will be performed. Participants will begin with their dominant hand and quickly move 9 cylindrical plastic pegs from a concave dish into 9 holes. Pegs will be placed in the holes 1 at a time and once all pegs are in a hole the participants will remove the pegs and return them to the dish. Each hand will be tested twice and the time of completion will be recorded with a handheld stop watch. The PASAT will be performed after the 9HPT to test cognitive function. This test consists of the playback of a series of pre-recorded numbers spoken on a computer. The participants are asked to add the last two spoken numbers which occur every three seconds for a 3 minute period of time. The number of correct answers is recorded by the test moderator.
5. Next the Isometric Strength of the knee extensors, knee flexors, plantar flexors, and dorsi-flexors will be measured. The participants will perform the strength tests from a seated position with the knee and hip joints at 90 degrees flexion. When testing ankle strength, the ankle will be at 90 degrees. Once participants are in the proper position they will be attached to a linear force transducer. Participants will slowly increase the force of the muscle group being tested for 3 sec from 0 to maximum. They will be instructed to produce maximum force for 3 seconds and then relax. Each muscle group will be tested at minimum 3 times. Testing will end when either there is a decrease in force between the last 2 trials performed or the force produced is less than 5% of the previous trial.
6. Once a month the investigators will visit each participant at their home. Prior to the visit, the participant will inform the investigators about the timing of their smoking to ensure that the blood draw with sodium heparin will occur no later than 15 min after smoking to ensure measurable THC, THC metabolites, CBD and CBN (cannabinol) levels. Blood THC, CBD and CBN content, along with THC phase I metabolites 11-OH-THC (active 11-hydroxy-THC) and THC-COOH (inactive 11-nor-9- carboxy-THC) will be determined using liquid chromatography-mass spectrometry in the Department of Chemistry under the direction of Dr. Denef. These values will inform on the participant's blood cannabinoid profile and the relative contents of non-psychoactive CBD and CBN versus psychoactive THC and its metabolites. Importantly, at each home session, participants will be asked about adverse effects and allergies related to marijuana.

PRE-POST ASSESSMENTS:

A Dual-Energy X-Ray Absorptiometry scan will be performed to assess body composition before and during the last month of the 3-month intervention for a total of 2 scans. Furthermore, participants will be asked to wear an ActiGraph accelerometer for 7 days to measure physical activity before and during the last month of the intervention. During non-wear times, participants will be asked to write any activities performed in a log.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with MS
* Age range 21-74 years of age
* Moderate disability (Patient Determined Disease Steps score 2-6)
* All participants must have a medical (red) card for medical marijuana use to treat their MS symptoms (such as neuropathic pain and spasticity), or currently be in the process of applying for a red card and be able to provide the prescription from their doctor.

Exclusion Criteria:

* Previous use of marijuana
* A relapse of disease symptoms in the last 60 days
* A condition unrelated to MS that would exacerbate fatigue, such as anemia, hypothyroidism, shiftwork-related fatigue, B12 deficiency, major sleep disorder, or major depressive disorder
* Medical diagnosis or condition that makes participating in exercise training dangerous, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than treated basal cell cancer), other neurological disorders
* History of heart attack or current diagnosis of cardiovascular disease
* History of seizure disorders (or on medications known to lower seizure threshold), hydrocephalus (buildup of fluid in the brain), or diabetes
* Alcohol dependence or abuse (>2 drinks/day), or present history (last six months) of drug abuse
* History of significant traumatic brain injury or hydrocephalus
* Pregnancy
* Recent hospitalization (within the last 3 months) or enforced bed rest/sedentary state
* Current participation in another research study that involves experiments on drugs or interventions which may influence motor and cognitive function.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Leg Strength | 1 year
  kg
Fatigue Severity Scale | 1 year
  Numeric Scale
25 foot walk test | 1 year
  Time (min)
9 hole peg test | 1 year
  Time (sec)
Paced Auditory Serial Addition Test | 1 year
  Time (min)
Becks Depression Inventory | 1 year
  Numeric Scale
Quality of Life | 1 year
  Numeric Scale
Pain Effect Scale. | 1 year
  Numeric Scale

SECONDARY OUTCOMES:
Fat Mass | 1 year
  kg
Lean Body Mass | 1 year
  kg

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, PhD, Principal Investigator — Colorado State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etemadi Y. Dual task cost of cognition is related to fall risk in patients with multiple sclerosis: a prospective study. Clin Rehabil. 2017 Feb;31(2):278-284. doi: 10.1177/0269215516637201. Epub 2016 Jul 10. PMID 26951347
- [Background] Ghanavati T, Salavati M, Karimi N, Negahban H, Ebrahimi Takamjani I, Mehravar M, Hessam M. Intra-limb coordination while walking is affected by cognitive load and walking speed. J Biomech. 2014 Jul 18;47(10):2300-5. doi: 10.1016/j.jbiomech.2014.04.038. Epub 2014 May 9. PMID 24861632
- [Background] Hart CL, Ilan AB, Gevins A, Gunderson EW, Role K, Colley J, Foltin RW. Neurophysiological and cognitive effects of smoked marijuana in frequent users. Pharmacol Biochem Behav. 2010 Sep;96(3):333-41. doi: 10.1016/j.pbb.2010.06.003. Epub 2010 Jun 18. PMID 20600251